CLINICAL TRIAL: NCT07359599
Title: A Randomized, Double-blind, Placebo-controlled, Multicentre Trial, Assessing the Impact of Ferric Carboxymaltose on Exercise Capacity and Functional Status in Pulmonary Hypertension
Brief Title: The Impact of IV Iron on Exercise Capacity and Quality of Life in Pulmonary Hypertension
Acronym: IRON-PH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: Federal Knowledge Centre (KCE) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Z-2025090; 2025-522936-14-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-09; First posted 2026-01-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Hypertension; Iron Deficiency
MeSH Terms: conditions — Hypertension, Pulmonary; Iron Deficiencies | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferric carboxymaltose (Experimental)
  Interventions: Drug: Ferric Carboxymaltose (FCM)
- Placebo (Placebo Comparator)
  Interventions: Drug: Sodium Chloride (NaCl) 0.9 %

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM) — Ferric Carboxymaltose (FCM), dosing and administration according to SmPC guidelines
  Arms: Ferric carboxymaltose
Drug: Sodium Chloride (NaCl) 0.9 % — Placebo, dosing and administration according to SmPC guidelines
  Arms: Placebo

SUMMARY:
Pulmonary hypertension (PH) is a condition characterized by elevated blood pressure in the pulmonary arteries. This leads to symptoms such as shortness of breath and a significantly reduced exercise capacity, resulting in a very poor quality of life. Currently, treatment options for PH are limited.

More than 60% of patients with PH develop iron deficiency. Studies have shown that this deficiency is associated with more severe symptoms, reduced exercise capacity, and even lower quality of life. Oral iron supplements are often ineffective in these patients due to impaired absorption in the intestines, caused by chronic low-grade inflammation-a common feature in PH.

Intravenous iron administration can rapidly correct the deficiency, but it remains unclear whether this also leads to clinical improvements such as enhanced exercise capacity, reduced shortness of breath, and improved quality of life. Moreover, the cost-effectiveness of this treatment is still unknown. The IRON-PH study aims to answer these questions.

As part of the IRON-PH study, 306 patients with pulmonary hypertension will be enrolled. Each patient will be randomized to receive either intravenous iron (ferric carboxymaltose) or intravenous placebo (NaCl 0.9%).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* WHO functional class II - IV
* Iron deficiency defined as TSAT <21% (no more than ≥3 months old at randomization)
* PH defined by echocardiography and/or right heart catheterization (RHC) according to the following WHO groups:

  * Group 1 PH:

    * Patients with a diagnosis of idiopathic PAH, hereditary PAH, drug induced PAH or PAH and associated with CTD or CHD (historical RHC available) on stable and optimized doses of PAH targeted therapies for at least 4 weeks before randomization.
    * Echocardiographic evidence of a high or intermediate probability for PH as per 2022 ESC PH guidelines.
  * Group 2 PH and baseline LVEF > 50% on imaging modality within last 6 months before randomization and on stable doses of loop diuretics and HFpEF therapies for 4 weeks. Group 2 PH can be included based on echocardiography or RHC.:

    * Echocardiography (<6mo before randomization):

      * Presence of LVH or LA-enlargement
      * E/e' >15 (at rest or exercise)
      * TRVmax >2.8 m/s (at rest) or mPAP/CO>3 mHg/L/min (exercise) or echocardiographic evidence of high or intermediate probability for PH as per 2022 ESC PH guidelines.
    * RHC (<6mo before randomization)

      * mPAP > 20 mmHg
      * PCWP > 15 mmHg at rest or PCWP/CO-slope > 2mmHg/L/min or exercise PCWP>25mmHg, or PCWP 13-15 mmHg with elevation ≥18mmHg after 500 cc Fluid Challenge
  * Group 4 PH:

    * Inoperable CTEPH
    * Persistent/recurrent CTEPH (> 1 year after endarterectomy or > 6 months after balloon pulmonary angioplasty) ineligible for balloon pulmonary angioplasty.
    * Echocardiographic evidence of a high or intermediate probability for PH as per 2022 ESC PH guidelines.

Exclusion Criteria:

* Screening haemoglobin < 8 g/dl or >15 g/dl
* Ferritin > 700 ng/mL
* Known hypersensitivity reaction to any component of FCM
* Group 1 PH associated with veno-occlusive diseases.
* Primary diagnosis of group 3 PH
* Primary diagnosis of group 5 PH
* Treatment with oral or other IV iron therapies at screening.
* Current or planned mechanical circulatory support or lung/heart transplantation.
* Any planned surgery or procedure leading to expected significant blood loss (defined as more than 250 ml = equal to 125mg of iron).
* Haemodialysis or peritoneal dialysis (current or planned within the next 24 weeks).
* Inability to return for follow up visits within the necessary windows
* Concurrently in a study with another investigational product.
* Uncorrected moderate to severe aortic stenosis (AVA <1.5cm² and mean gradient >20 mmHg) or severe valvular regurgitation (except tricuspid regurgitation)
* Impression by investigator that patient cannot perform a 6MWT
* Active infection as judged by the investigator.
* Pregnancy or desire to become pregnant during the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change in 6MWD | From baseline to 24 week follow-up
  Change in 6-minute walking distance (6MWD) from baseline to 24 week follow-up

SECONDARY OUTCOMES:
Change in MLHFQ | Baseline to 24 week follow-up
  Change in Minnesota Living with Heart Failure Questionnaire (MLHFQ) score from baseline to 24 week follow-up.
  Total Score: Sum of all 21 items (0-105) Higher Score = Worse QoL: A higher number indicates a greater negative impact from heart failure Lower Score = Better QoL: A lower score suggests less limitation
Change in EQ5D5L | Baseline to 24 week follow-up
  Change in EuroQol 5 dimensions - 5 levels questionnaire score from baseline to 24 week follow-up EQ-5D-5L combiines responses from five health dimensions, each with five severity levels to create a 5-digit health state code, then applying country-specific "value sets" (valuation matrices) to convert this code into a single Index Score (Utility Score), ranging from <0 (worst) to 1 (best health), plus a separate EQ-VAS score (0-100) for overall self-rated health.
  Dimensions: Mobility, self-care, usual activities, pain/discomfort, anxiey/depression Levels: 1 no problem, 2 slight problems, 3 moderate problems, 4 severe problems, 5 unable to/extreme problems Example of 5-digit state code: 12345 indicates no problems with mobility, slight problems with self-care, moderate problems with usual activities, severe pain/discomfort and extreme anxiety/depression
Change in FSS | Baseline to 24 week follow-up
  Change in Fatigue Severity Scale (FSS) score from baseline to 24 weeks Total score: sum of all scores (ranging between 9 - 63) Higher Scores = More Fatigue Lower Scores = Less Fatigue
Developing composite clinical worsening event | From first patient Day 1 (Baseline) to study completion, an average of 2 years
  The hazard ratio between treatment arms in developing the composite clinical worsening event in the overall trial population

CONTACTS AND LOCATIONS:
Locations (7):
- Belgium (7):
  - AZORG, Aalst
  - Hôpital Erasme, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHU Charleroi-Chimay, Lodelinsart
  - CHU UCL Namur, Yvoir

IPD SHARING:
Plan to Share IPD: No